

# Statistical Analysis Plan

A prospective international multicentre randomized, double-blind, placebo-controlled parallel-group clinical trial to evaluate the safety and efficacy of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in their sequential use in patients in the acute and early recovery periods of ischaemic stroke (MIR)

NCT Number: NCT06437626

Pharmasoft

November 12, 2021



# Plan of statistical analysis of efficacy and safety parameters version 1.0 dated 12.11.2021 based on the results of

"A prospective international multicentre randomized double-blind placebocontrolled parallel-group clinical trial to evaluate the safety and efficacy of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in their sequential use in patients in the acute and early recovery periods of ischaemic stroke (IS)" under protocol #PHS-APIS-004-MEX-SOL-TAB, version 1.3 dated 07.06.2021.



Approval sheet for the statistical analysis of efficacy and safety parameters, version 1.0 dated 12.11.2021, in "Prospective international multicentre randomized double-blind placebo-controlled parallel-group clinical trial to evaluate the safety and efficacy of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in their sequential use in patients in the acute and early recovery periods of ischaemic stroke (IS)", protocol #PHS-APIS-004-MEX-SOL-TAB, version 1.3 dated 07.06.2021.

| Project Manager | | |
|-------------------------------------------|-----------|------------|
| Balandin M.O. | (signed) | 07.06.2021 |
| FULL NAME | signature | date |
| Statistician: | | |
| Volin A.Y. | (signed) | 07.06.2021 |
| FULL NAME | signature | date |
| Responsible Person on the Sponsor's side: | | |
| Chizhova G.A. | (signed) | 07.06.2021 |
| FULL NAME | signature | date |



# History of changes to the document

| Version number Date of issue | Data of issue | Amendments |
|------------------------------|----------------------------|--------------|
| | Section Modifications made | |
| 1.0 | 12.11 .2021 | New document |



# **Table of Contents**

| 1. | Trial background | 9 |
|---|---|---|
| 2. | Purpose of data statistical analysis | 11 |
| 3. | Deviations from protocol | 12 |
| 4. | Trial procedures | 13 |
| 5. | Randomization | 13 |
| 6. | Main and additional trial parameters to be assessed in the course of the trial | 26 |
| 7. | Statistical hypothesis | 27 |
| 8. | Estimation of the required sample size | 28 |
| 9. | Statistical evaluation of efficacy parameters and pharmacodynamic effects | 29 |
| 10. | Safety analysis | 30 |
| 11. | Patient populations to be analysed | 33 |
| 12. | Interim analysis | 34 |
| 13. | Table templates | 34 |



# List of tables

| Table 1. Randomization scheme developed by Smooth Drug Development | . 13 |
|---|---|
| Table 2. Results of assessment of normality of distribution of indicators (template) | . 34 |
| Table 3. Statistical analysis of the primary endpoint (template) | . 42 |
| Table 4. Outcome of primary endpoint analysis (template) | . 42 |
| Table 5. Statistical analysis of the NIHSS scale (template) | . 43 |
| Table 6. Statistical analysis of secondary endpoints (quantitative data, template) | . 44 |
| Table 7. Statistical analysis of pharmacodynamic effect indicators (template) | |
| Table 8. Statistical analysis of the proportion of disabled patients (template) | . 46 |
| Table 9. Statistical analysis of safety indicators (quantitative data, template) | . 46 |
| Table 10. Statistical analysis of vital signs (quantitative data, template) | . 46 |
| Table 11. Safety performance assessment results: repeated measures analysis of variance | |
| (template) | . 47 |
| Table 12. Results of safety indicators assessment: non-parametric repeated measures analyst | is |
| of variance (Friedman test, template) | |
| Table 13. Frequency analysis of safety performance outcome assessment (template) | . 48 |
| Table 14. Frequency analysis of the safety outcome measure score (clinical significance, | |
| template) | . 48 |
| Table 15. Statistical analysis of ECG (template) | . 49 |
| Table 16. Statistical analysis of physical examination parameters (outcome measure, | |
| template) | . 49 |
| Table 17. Distribution of patients by ender (template) | |
| Table 18. Baseline patient characteristics (template) | |
| Table 19. Total number of AEs (template) | |
| Table 20. Relative risk of AEs (template) | |
| Table 21. Analysing the distribution of AEs by severity (template) | |
| Table 22. Relationship of AEs to investigational drug (template) | |
| Table 23: Analysis of the distribution of AEs by drug administration (template) | |
| Table 24. Analysis of the distribution of AEs by foreseeability (template) | |
| Table 25. Analysis of AR distribution (template) | |
| Table 26. Analysis of the distribution of AEs by seriousness (template) | |
| Table 27. Analysing the distribution of AEs by actions taken (template) | |
| Table 28. Analysis of the distribution of AEs by outcome (template) | |
| Table 29. Summary table of the incidence of reported AEs in the group taking Mexidol by | |
| severity with randomization numbers of patients (N=) (template) | . 54 |
| Table 30. Summary table of the incidence of reported AEs in the group taking placebo by | |
| severity with randomization numbers of patients (N=) (template) | . 54 |
| Table 31. Summary table of the incidence of AEs after taking each drug (template) | |
| Table 32. List of all adverse events for each patient (template) | |
| Table 33. MedDRA version classification of AEs (template) | |
| Table 34. Summary table of the incidence of reported SAEs in the group taking Mexidol by | |
| severity with randomization numbers of patients (N=) (template) | . 56 |
| Table 35. Summary table of the incidence of reported SAEs in the placebo group by grade | _ |
| with randomization numbers of patients (N=) (template) | . 56 |





| Table 36. Summ | nary table of the incidence of SAEs after taking each drug (template) | 56 |
|---|---|---|
| Table 37. List of | of all serious adverse events for each patient (template) | 57 |
| Table 38. MedD | ORA version classification of SAEs (template) | 57 |



#### List of abbreviations

ALT - alanine aminotransferase:

AST - aspartate aminotransferase;

DBP - diastolic blood pressure;

IV - intravenous:

IM - intramuscular;

GGTP - gamma-glutamyl transpeptidase;

CI - confidence interval;

BMI - Body Mass Index;

MP - medicinal product;

AE - Adverse event;

AR - adverse reaction;

SBD - systolic blood pressure;

SAE - serious adverse event;

HR - respiratory rate;

HR - Heart rate;

ALP - alkaline phosphatase;

eCRF - electronic case report form;

ECG - electrocardiography.

ANOVA - Analysis of variance;

CTCAE - Common Toxicity Criteria for Adverse Events;

GCP - Good Clinical Practice;

HADS - Hospital Anxiety and Depression Scale;

ITT - Intent-to-treat population, includes all randomized patients regardless of investigational product/placebo administration

MedDRA - Medical Dictionary for Regulatory Activities;

mITT - modified Intent-to-treat population includes patients who have completed the full course of therapy, regardless of the presence of violations/ deviations from the Protocol;

MoCA - Montreal Cognitive Assessment Scale;

mRS - Modified Rankin Scale:

NIHSS - National Institutes of Health Stroke Scale;

PP - Per protocol population includes patients who completed the trial according to the Protocol. In the tables of efficacy and safety of the medicinal products Mexidol® solution for intravenous and intramuscular injection, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) vs. placebo the following parameters of descriptive statistics will be given:

N - number of valid observations;

Mean - arithmetic mean;

Median - middle point in a dataset

Min - minimum value:

Max - maximum value;

Q<sub>1</sub> - lower quartile;

Q<sub>3</sub> - upper quartile;

Version 1.0 of 12.11.2021

Protocol-Specific Version for Protocol #PHS-

APIS-004-MEX-SOL-TAV. version 1.3 dated

07.06.2021

**CONFIDENTIAL** 



SD - standard deviation;

CV - coefficient of variation.

#### 1. Trial background

**Trial title:** Prospective international multicentre randomized, double-blind, placebocontrolled, parallel-group clinical trial to evaluate the safety and efficacy of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC Pharmasoft LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in their sequential use in patients in the acute and early recovery periods of ischaemic stroke (MIR).

Protocol No.: PHS-APIS-004-MEX-SOL-TAB, version 1.3 dated 07.06.2021

Sponsor: RPC PHARMASOFT LLC, Russia

**Investigational product:** Mexidol® solution for intravenous and intramuscular injection, 50 mg/ml (RPC PHARMASOFT LLC, Russia) 10 ml (500 mg) BID by intravenous drip in 100-200 ml of 0.9% NaCl solution for 10 days and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) 1 tablet TID for the next 60 days.

**Comparison product:** Placebo 1, solution for intravenous and intramuscular injection, 10 ml BID by intravenous drip in 100-200 ml of 0.9% NaCl solution for 10 days and Placebo 2, film-coated tablets, 1 tablet TID for the next 60 days.

**Development Phase: III** 

**Trial design:** A prospective multicentre, randomized, double-blind, parallel-group comparative clinical trial.

Number of patients: 304

**Purpose of the trial:** comparative evaluation of efficacy and safety of therapy with Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in comparison with placebo during their sequential use in patients in the acute and early recovery periods of ischaemic stroke.

#### **Trial objectives:**

- 1. To evaluate the efficacy of Mexidol® solution for intravenous and intramuscular injection, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) during their sequential use in patients in the acute and early recovery periods of ischaemic stroke vs. placebo.
- 2. To carry out a comparative evaluation of the frequency and severity of adverse events of Mexidol® solution for intravenous and intramuscular injection, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) during their sequential use in patients in the acute and early recovery periods of ischaemic stroke vs. placebo.

Additional objective: To carry out a comparative evaluation of pharmacodynamic effects of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) during their sequential use in patients in the acute and early recovery periods of ischaemic stroke vs. placebo.



#### **Primary endpoint:**

The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the end of therapy vs. baseline (in scores).

#### **Secondary endpoints:**

- 1. The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the end of parenteral therapy vs. baseline (in scores).
- 2. Proportion of disabled patients (mRS score 3 or more) at the end of therapy vs. baseline;
- 3. Proportion of disabled patients (mRS score 3 or more) at the end of parenteral therapy vs. baseline;
- 4. The magnitude of change in the patient's NIHSS (National Institutes of Health Stroke Scale) score at the end of therapy vs. baseline (in scores).
- 5. The magnitude of change in the patient's NIHSS (National Institutes of Health Stroke Scale) score at the end of parenteral therapy vs. baseline (in scores).
- 6. The magnitude of change in the patient's MoCA cognitive status score at the end of therapy vs. baseline (in scores).
- 7. The magnitude of change in the patient's MoCA cognitive status score at the end of parenteral therapy vs. baseline (in scores).
- 8. The magnitude of change in the patient's Rivermead Mobility Index score at the end of therapy vs. baseline (in scores).
- 9. The magnitude of change in the results of the patient's state assessment by the Rivermead mobility index at the end of the parenteral course of therapy vs. baseline (in scores).
- 10. The magnitude of change in the patient's HADS score at the end of therapy vs. baseline (in scores).
- 11. The magnitude of change in the patient's HADS score at the end of parenteral therapy vs. baseline (in scores).

#### Criteria for assessing pharmacodynamic effects:

- 1. The magnitude of change in the results of assessment of LPO activity (malonic dialdehyde) and AOS indicators (superoxide dismutase, Se-dependent glutathione peroxidase) at the end of therapy vs. baseline;
- 2. The magnitude of change in the results of assessment of LPO activity (malonic dialdehyde) and AOS indicators (superoxide dismutase, Se-dependent glutathione peroxidase) at the end of the parenteral course of therapy vs. baseline;
- 3. The magnitude of change in the results of evaluation of laboratory parameters reflecting ED (Willebrandt factor, endothelin 1, homocysteine) and antihypoxant effect (hypoxia-inducible factor HIF-I $\alpha$ , lactate, neuron-specific enolase) at the end of therapy vs. baseline:
- 4. The magnitude of change in the results of evaluation of laboratory parameters reflecting ED (Willebrandt factor, endothelin 1, homocysteine) and antihypoxant effect (hypoxia-inducible factor HIF-1 $\alpha$ , lactate, neuron-specific enolase) at the end of the parenteral course of therapy vs. baseline.



# **Safety parameters**

Safety and tolerability will be assessed throughout the trial (from first use of the investigational product/placebo) using the following data:

- 1. AE/SAE reports data,
- 2. Physical examination data, vital signs (BP, HR, respiratory rate, body temperature),
- 3. Indicators of laboratory analyses and instrumental methods of examination.

A conclusion on the safety of the investigational product will be made after statistical evaluation of all AEs, including serious SAEs with at least a possible association with the use of the investigational product.

**Applicable significance level:** probability of a 1st kind of error is set at 5%. As an interim analysis of the primary endpoint data is planned, a genus I error correction approach  $\alpha$  ( $\alpha$  = 0.0294) will be used to prove the hypothesis of "superiority" of investigational product therapy vs. placebo therapy for the primary efficacy criterion.

## 2. Purpose of data statistical analysis

The purpose of the development of this Statistical Analysis Plan is to describe the planned analysis of efficacy and safety data in the "Prospective international multicentre randomized double-blind placebo-controlled parallel-group clinical trial to evaluate the efficacy and safety of Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) in their sequential use in patients in the acute and early recovery periods of ischaemic stroke (IS)" under protocol #PHS-APIS-004-MEX-SOL-TAB, version 1.3 dated 07.06.2021, for inclusion of the results in the Clinical Trial Report.

The results obtained according to the planned statistical analysis of the data presented in this document will be used in the submission of the registration dossier for the drug to the regulatory authorities, as well as in the writing of publications on the materials of the conducted clinical trial.

The trial will be conducted in accordance with the Protocol, in strict compliance with applicable regulatory requirements, including but not limited to:

- Constitution of the Russian Federation:
- Current version of the Federal Law of the Russian Federation dated 21 November 2011 No. 323-FZ "On the Fundamentals of Health Protection of Citizens in the Russian Federation";
- Current version of the Federal Law of the Russian Federation No. 61-FZ "On Circulation of Medicines" dated 12 April 2010;
- Current version of the Federal Law of the Russian Federation dated 27 July 2006 N 152-FZ "On Personal Data"
- Order of the Ministry of Health of the Russian Federation No. 200 n of 01.04.2016. "On Approval of the Rules of Good Clinical Practice";
- Russian National Standard GOST R 52379-2005 "Good Clinical Practice", which complies with the standards of the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceutical Products for Human Use (ICH) Good Clinical Practice Guidelines (ICH-GCP);



- Rules of Good Clinical Practice of the Eurasian Economic Union, approved by the Decision of the Council of the Eurasian Economic Commission dated 3 November 2016 No. 79:
- Rules of Compulsory Life and Health Insurance for Patients Participating in Clinical studies of a Medicinal Product approved by Resolution of the Government of the Russian Federation No. 714 dated 13 September 2010;
- Resolution of the Government of the Russian Federation No. 393 dated 18 May 2011
   "On Amendments to the Model Rules for Compulsory Life and Health Insurance for Patients Participating in Clinical studies of a Medicinal Product";
- Rules of the International Conference on Harmonisation of Technical Requirements for Registration of Medicinal Products for Human Use;
- The World Medical Association's 1964 Declaration of Helsinki, most recently revised (Fortaleza, 2013);
- Guidelines for Expertise of Medicinal Products of FGBU NCESMP of the Ministry of Health of Russia (Moscow, 2013)
- Order of the Federal Service for Healthcare Oversight No. 1071 dated 15.02.2017 "On Approval of the Procedure for Pharmacovigilance";
- Order of the Ministry of Health and Social Development of the Russian Federation No. 757n dated 26.08.2010 "On Approval of the Procedure for Monitoring the Safety of Medicinal Products for Medical Use, Registration of Adverse Actions, Serious Adverse Reactions, Unexpected Adverse Reactions in the Use of Medicinal Products for Medical Use":

Statistical evaluation of efficacy and safety parameters will be performed in accordance with the Drug Evaluation Guidelines (Volume I. - FGBU NCESMP, Moscow, 2014), Guidelines on the principles of application of biostatistics in clinical trials of medicinal products (Annex to the recommendation of the EEC Collegium from 03.11.2020 No. 2014) and general recommendations on biomedical statistics (ICH Topic E9 Statistical Principles for Clinical Trials, CPMP/ICH/363/96, 1998; Sergienko V.I., Bondareva I.B. Mathematical Statistics in Clinical Trials, Moscow: GEOSTAR-Media, 2006).

# 3. Deviations from protocol

A statistical plan has been prepared and will be agreed prior to the statistical analysis. Statistical analyses were planned according to the Clinical Trial Protocol. Deviations from the protocol in statistical analyses are not planned. Any deviation from the protocol is permitted only in an emergency or after written authorization from the Sponsor. If there is a deviation from the planned statistical analysis, all changes will be identified compared to the methods described in the statistical analysis plan. Similarly, if any additional changes are required after the analysis has been performed, this will be reflected in the Clinical Trial Report. All deviations of the present from the statistical analysis plan with their justification will be reported in the Clinical Trial Report. No changes will be made to the list of parameters to be evaluated. Statistical analysis methods may be changed if this would facilitate a more correct and informative analysis, any changes will be described and justified in the final Clinical Trial Report.



# 4. Trial procedures



#### 5. Randomization

Table 1. Randomization scheme developed by Smooth Drug Development

| Country | Block number | Randomization code | Therapy |
|------------------------|--------------|--------------------|---------|
| Republic of Kazakhstan | 001 | 616 | В |
| Republic of Kazakhstan | 001 | 174 | A |
| Republic of Kazakhstan | 001 | 637 | В |
| Republic of Kazakhstan | 001 | 869 | A |
| Republic of Kazakhstan | 2 | 455 | A |
| Republic of Kazakhstan | 2 | 548 | В |
| Republic of Kazakhstan | 2 | 687 | A |
| Republic of Kazakhstan | 2 | 809 | В |
| Republic of Kazakhstan | 3 | 810 | В |
| Republic of Kazakhstan | 3 | 680 | A |
| Republic of Kazakhstan | 3 | 294 | A |
| Republic of Kazakhstan | 3 | 513 | В |
| Republic of Kazakhstan | 4 | 180 | A |
| Republic of Kazakhstan | 4 | 467 | В |
| Republic of Kazakhstan | 4 | 986 | A |
| Republic of Kazakhstan | 4 | 365 | В |
| Republic of Kazakhstan | 5 | 865 | A |
| Republic of Kazakhstan | 5 | 678 | В |
| Republic of Kazakhstan | 5 | 671 | В |
| Republic of Kazakhstan | 5 | 677 | A |




| Country | Block number | Randomization code | Therapy |
|------------------------|--------------|--------------------|---------|
| Republic of Uzbekistan | 6 | 641 | В |
| Republic of Uzbekistan | 6 | 214 | A |
| Republic of Uzbekistan | 6 | 189 | A |
| Republic of Uzbekistan | 6 | 223 | В |
| Republic of Uzbekistan | 7 | 611 | A |
| Republic of Uzbekistan | 7 | 450 | В |
| Republic of Uzbekistan | 7 | 213 | В |
| Republic of Uzbekistan | 7 | 688 | A |
| Republic of Uzbekistan | 8 | 498 | В |
| Republic of Uzbekistan | 8 | 427 | A |
| Republic of Uzbekistan | 8 | 217 | В |
| Republic of Uzbekistan | 8 | 505 | A |
| Republic of Uzbekistan | 9 | 315 | В |
| Republic of Uzbekistan | 9 | 411 | A |
| Republic of Uzbekistan | 9 | 699 | В |
| Republic of Uzbekistan | 9 | 626 | A |
| Republic of Uzbekistan | 10 | 330 | A |
| Republic of Uzbekistan | 10 | 983 | В |
| Republic of Uzbekistan | 10 | 249 | В |
| Republic of Uzbekistan | 10 | 566 | A |
| Russian Federation | 11 | 933 | В |
| Russian Federation | 11 | 393 | A |
| Russian Federation | 11 | 507 | В |
| Russian Federation | 11 | 493 | A |
| Russian Federation | 12 | 524 | A |
| Russian Federation | 12 | 648 | В |
| Russian Federation | 12 | 697 | A |
| Russian Federation | 12 | 912 | В |
| Russian Federation | 13 | 303 | A |
| Russian Federation | 13 | 228 | В |
| Russian Federation | 13 | 802 | A |
| Russian Federation | 13 | 738 | В |
| Russian Federation | 14 | 435 | A |
| Russian Federation | 14 | 732 | В |
| Russian Federation | 14 | 456 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 14 | 279 | В |
| Russian Federation | 15 | 394 | В |
| Russian Federation | 15 | 804 | A |
| Russian Federation | 15 | 274 | A |
| Russian Federation | 15 | 238 | В |
| Russian Federation | 16 | 285 | A |
| Russian Federation | 16 | 160 | В |
| Russian Federation | 16 | 170 | В |
| Russian Federation | 16 | 876 | A |
| Russian Federation | 17 | 846 | В |
| Russian Federation | 017 | 757 | A |
| Russian Federation | 017 | 555 | A |
| Russian Federation | 017 | 131 | В |
| Russian Federation | 018 | 700 | A |
| Russian Federation | 018 | 154 | В |
| Russian Federation | 018 | 132 | В |
| Russian Federation | 018 | 197 | A |
| Russian Federation | 019 | 235 | A |
| Russian Federation | 019 | 835 | В |
| Russian Federation | 019 | 818 | В |
| Russian Federation | 019 | 656 | A |
| Russian Federation | 020 | 291 | В |
| Russian Federation | 020 | 337 | A |
| Russian Federation | 020 | 151 | В |
| Russian Federation | 020 | 785 | A |
| Russian Federation | 21 | 608 | В |
| Russian Federation | 21 | 344 | A |
| Russian Federation | 21 | 770 | В |
| Russian Federation | 21 | 772 | A |
| Russian Federation | 022 | 936 | В |
| Russian Federation | 022 | 923 | A |
| Russian Federation | 022 | 758 | A |
| Russian Federation | 022 | 705 | В |
| Russian Federation | 023 | 902 | A |
| Russian Federation | 023 | 329 | В |


07.06.2021

Protocol-Specific Version for Protocol #PHS-APIS-004-MEX-SOL-TAV. version 1.3 dated

CONFIDENTIAL

page 15 of 58



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 023 | 198 | A |
| Russian Federation | 023 | 728 | В |
| Russian Federation | 024 | 156 | A |
| Russian Federation | 024 | 402 | В |
| Russian Federation | 024 | 459 | В |
| Russian Federation | 024 | 193 | A |
| Russian Federation | 025 | 999 | В |
| Russian Federation | 025 | 252 | A |
| Russian Federation | 025 | 900 | В |
| Russian Federation | 025 | 306 | A |
| Russian Federation | 026 | 874 | В |
| Russian Federation | 026 | 305 | A |
| Russian Federation | 026 | 173 | В |
| Russian Federation | 026 | 470 | A |
| Russian Federation | 027 | 251 | A |
| Russian Federation | 027 | 155 | В |
| Russian Federation | 027 | 119 | В |
| Russian Federation | 027 | 652 | A |
| Russian Federation | 028 | 613 | В |
| Russian Federation | 028 | 929 | A |
| Russian Federation | 028 | 896 | A |
| Russian Federation | 028 | 492 | В |
| Russian Federation | 029 | 623 | A |
| Russian Federation | 029 | 984 | В |
| Russian Federation | 029 | 761 | A |
| Russian Federation | 029 | 568 | В |
| Russian Federation | 030 | 917 | A |
| Russian Federation | 030 | 599 | В |
| Russian Federation | 030 | 601 | В |
| Russian Federation | 030 | 488 | A |
| Russian Federation | 031 | 447 | В |
| Russian Federation | 031 | 260 | A |
| Russian Federation | 031 | 750 | A |
| Russian Federation | 031 | 877 | В |
| Russian Federation | 032 | 694 | В |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 032 | 169 | A |
| Russian Federation | 032 | 509 | A |
| Russian Federation | 032 | 273 | В |
| Russian Federation | 033 | 428 | A |
| Russian Federation | 033 | 144 | В |
| Russian Federation | 033 | 192 | В |
| Russian Federation | 033 | 469 | A |
| Russian Federation | 034 | 922 | В |
| Russian Federation | 034 | 893 | A |
| Russian Federation | 034 | 253 | В |
| Russian Federation | 034 | 817 | A |
| Russian Federation | 035 | 242 | В |
| Russian Federation | 035 | 811 | A |
| Russian Federation | 035 | 130 | В |
| Russian Federation | 035 | 711 | A |
| Russian Federation | 036 | 609 | В |
| Russian Federation | 036 | 476 | A |
| Russian Federation | 036 | 219 | В |
| Russian Federation | 036 | 395 | A |
| Russian Federation | 037 | 484 | В |
| Russian Federation | 037 | 718 | A |
| Russian Federation | 037 | 290 | A |
| Russian Federation | 037 | 152 | В |
| Russian Federation | 038 | 300 | A |
| Russian Federation | 038 | 992 | В |
| Russian Federation | 038 | 840 | В |
| Russian Federation | 038 | 230 | A |
| Russian Federation | 039 | 985 | В |
| Russian Federation | 039 | 946 | A |
| Russian Federation | 039 | 769 | A |
| Russian Federation | 039 | 522 | В |
| Russian Federation | 040 | 736 | В |
| Russian Federation | 040 | 808 | A |
| Russian Federation | 040 | 431 | В |
| Russian Federation | 040 | 495 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 041 | 137 | В |
| Russian Federation | 041 | 970 | A |
| Russian Federation | 041 | 905 | A |
| Russian Federation | 041 | 715 | В |
| Russian Federation | 042 | 215 | A |
| Russian Federation | 042 | 508 | В |
| Russian Federation | 042 | 774 | A |
| Russian Federation | 042 | 832 | В |
| Russian Federation | 043 | 713 | A |
| Russian Federation | 043 | 782 | В |
| Russian Federation | 043 | 250 | В |
| Russian Federation | 043 | 432 | A |
| Russian Federation | 044 | 501 | В |
| Russian Federation | 044 | 845 | A |
| Russian Federation | 044 | 960 | A |
| Russian Federation | 044 | 667 | В |
| Russian Federation | 045 | 570 | В |
| Russian Federation | 045 | 903 | A |
| Russian Federation | 045 | 257 | В |
| Russian Federation | 045 | 943 | A |
| Russian Federation | 046 | 413 | В |
| Russian Federation | 046 | 857 | A |
| Russian Federation | 046 | 218 | A |
| Russian Federation | 046 | 825 | В |
| Russian Federation | 047 | 500 | A |
| Russian Federation | 047 | 650 | В |
| Russian Federation | 047 | 875 | A |
| Russian Federation | 047 | 849 | В |
| Russian Federation | 048 | 227 | В |
| Russian Federation | 048 | 976 | A |
| Russian Federation | 048 | 220 | A |
| Russian Federation | 048 | 165 | В |
| Russian Federation | 049 | 696 | В |
| Russian Federation | 049 | 379 | A |
| Russian Federation | 049 | 403 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 049 | 147 | В |
| Russian Federation | 050 | 582 | В |
| Russian Federation | 050 | 157 | A |
| Russian Federation | 050 | 539 | В |
| Russian Federation | 050 | 642 | A |
| Russian Federation | 051 | 831 | В |
| Russian Federation | 051 | 884 | A |
| Russian Federation | 051 | 504 | В |
| Russian Federation | 051 | 727 | A |
| Russian Federation | 052 | 270 | A |
| Russian Federation | 052 | 210 | В |
| Russian Federation | 052 | 895 | A |
| Russian Federation | 052 | 120 | В |
| Russian Federation | 053 | 102 | A |
| Russian Federation | 053 | 380 | В |
| Russian Federation | 053 | 239 | A |
| Russian Federation | 053 | 466 | В |
| Russian Federation | 054 | 624 | A |
| Russian Federation | 054 | 229 | В |
| Russian Federation | 054 | 996 | A |
| Russian Federation | 054 | 768 | В |
| Russian Federation | 055 | 815 | A |
| Russian Federation | 055 | 640 | В |
| Russian Federation | 055 | 339 | В |
| Russian Federation | 055 | 562 | A |
| Russian Federation | 056 | 887 | В |
| Russian Federation | 056 | 338 | A |
| Russian Federation | 056 | 378 | В |
| Russian Federation | 056 | 942 | A |
| Russian Federation | 057 | 867 | В |
| Russian Federation | 057 | 837 | A |
| Russian Federation | 057 | 918 | A |
| Russian Federation | 057 | 264 | В |
| Russian Federation | 058 | 232 | В |
| Russian Federation | 058 | 945 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 058 | 363 | В |
| Russian Federation | 058 | 627 | A |
| Russian Federation | 059 | 981 | A |
| Russian Federation | 059 | 353 | В |
| Russian Federation | 059 | 209 | В |
| Russian Federation | 059 | 112 | A |
| Russian Federation | 060 | 765 | В |
| Russian Federation | 060 | 256 | A |
| Russian Federation | 060 | 904 | В |
| Russian Federation | 060 | 163 | A |
| Russian Federation | 061 | 162 | A |
| Russian Federation | 061 | 779 | В |
| Russian Federation | 061 | 776 | A |
| Russian Federation | 061 | 939 | В |
| Russian Federation | 062 | 991 | В |
| Russian Federation | 062 | 263 | A |
| Russian Federation | 062 | 520 | A |
| Russian Federation | 062 | 325 | В |
| Russian Federation | 063 | 899 | A |
| Russian Federation | 063 | 590 | В |
| Russian Federation | 063 | 533 | В |
| Russian Federation | 063 | 327 | A |
| Russian Federation | 064 | 222 | A |
| Russian Federation | 064 | 592 | В |
| Russian Federation | 064 | 871 | В |
| Russian Federation | 064 | 168 | A |
| Russian Federation | 065 | 979 | В |
| Russian Federation | 065 | 659 | A |
| Russian Federation | 065 | 474 | A |
| Russian Federation | 065 | 299 | В |
| Russian Federation | 066 | 308 | A |
| Russian Federation | 066 | 587 | В |
| Russian Federation | 066 | 318 | В |
| Russian Federation | 066 | 407 | A |
| Russian Federation | 067 | 494 | В |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 067 | 527 | A |
| Russian Federation | 067 | 645 | В |
| Russian Federation | 067 | 212 | A |
| Russian Federation | 068 | 878 | В |
| Russian Federation | 068 | 658 | A |
| Russian Federation | 068 | 702 | В |
| Russian Federation | 068 | 812 | A |
| Russian Federation | 069 | 345 | В |
| Russian Federation | 069 | 361 | A |
| Russian Federation | 069 | 775 | В |
| Russian Federation | 069 | 201 | A |
| Russian Federation | 070 | 657 | A |
| Russian Federation | 070 | 397 | В |
| Russian Federation | 070 | 543 | A |
| Russian Federation | 070 | 401 | В |
| Russian Federation | 071 | 730 | В |
| Russian Federation | 071 | 343 | A |
| Russian Federation | 071 | 559 | A |
| Russian Federation | 071 | 980 | В |
| Russian Federation | 072 | 646 | A |
| Russian Federation | 072 | 418 | В |
| Russian Federation | 072 | 851 | В |
| Russian Federation | 072 | 261 | A |
| Russian Federation | 073 | 585 | В |
| Russian Federation | 073 | 506 | A |
| Russian Federation | 073 | 490 | A |
| Russian Federation | 073 | 692 | В |
| Russian Federation | 074 | 799 | В |
| Russian Federation | 074 | 489 | A |
| Russian Federation | 074 | 178 | В |
| Russian Federation | 074 | 243 | A |
| Russian Federation | 075 | 967 | В |
| Russian Federation | 075 | 673 | A |
| Russian Federation | 075 | 862 | В |
| Russian Federation | 075 | 346 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 076 | 630 | В |
| Russian Federation | 076 | 644 | A |
| Russian Federation | 076 | 436 | A |
| Russian Federation | 076 | 792 | В |
| Russian Federation | 077 | 963 | В |
| Russian Federation | 077 | 240 | A |
| Russian Federation | 077 | 689 | A |
| Russian Federation | 077 | 150 | В |
| Russian Federation | 078 | 265 | В |
| Russian Federation | 078 | 433 | A |
| Russian Federation | 078 | 451 | В |
| Russian Federation | 078 | 534 | A |
| Russian Federation | 079 | 948 | В |
| Russian Federation | 079 | 940 | A |
| Russian Federation | 079 | 564 | В |
| Russian Federation | 079 | 858 | A |
| Russian Federation | 080 | 183 | A |
| Russian Federation | 080 | 479 | В |
| Russian Federation | 080 | 485 | В |
| Russian Federation | 080 | 748 | A |
| Russian Federation | 081 | 384 | A |
| Russian Federation | 081 | 586 | В |
| Russian Federation | 081 | 575 | A |
| Russian Federation | 081 | 368 | В |
| Russian Federation | 082 | 593 | В |
| Russian Federation | 082 | 883 | A |
| Russian Federation | 082 | 916 | A |
| Russian Federation | 082 | 224 | В |
| Russian Federation | 083 | 944 | В |
| Russian Federation | 083 | 990 | A |
| Russian Federation | 083 | 625 | A |
| Russian Federation | 083 | 952 | В |
| Russian Federation | 084 | 499 | A |
| Russian Federation | 084 | 108 | В |
| Russian Federation | 084 | 698 | В |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 084 | 607 | A |
| Russian Federation | 085 | 675 | A |
| Russian Federation | 085 | 733 | В |
| Russian Federation | 085 | 669 | A |
| Russian Federation | 085 | 783 | В |
| Russian Federation | 086 | 679 | A |
| Russian Federation | 086 | 472 | В |
| Russian Federation | 086 | 115 | A |
| Russian Federation | 086 | 597 | В |
| Russian Federation | 087 | 289 | В |
| Russian Federation | 087 | 726 | A |
| Russian Federation | 087 | 594 | A |
| Russian Federation | 087 | 313 | В |
| Russian Federation | 088 | 563 | A |
| Russian Federation | 088 | 268 | В |
| Russian Federation | 088 | 710 | В |
| Russian Federation | 088 | 124 | A |
| Russian Federation | 089 | 158 | В |
| Russian Federation | 089 | 376 | A |
| Russian Federation | 089 | 387 | В |
| Russian Federation | 089 | 388 | A |
| Russian Federation | 090 | 856 | A |
| Russian Federation | 090 | 237 | В |
| Russian Federation | 090 | 879 | A |
| Russian Federation | 090 | 236 | В |
| Russian Federation | 091 | 182 | A |
| Russian Federation | 091 | 629 | В |
| Russian Federation | 091 | 889 | В |
| Russian Federation | 091 | 558 | A |
| Russian Federation | 092 | 719 | A |
| Russian Federation | 092 | 553 | В |
| Russian Federation | 092 | 245 | В |
| Russian Federation | 092 | 292 | A |
| Russian Federation | 093 | 414 | В |
| Russian Federation | 093 | 618 | A |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 093 | 516 | A |
| Russian Federation | 093 | 781 | В |
| Russian Federation | 094 | 544 | В |
| Russian Federation | 094 | 880 | A |
| Russian Federation | 094 | 763 | В |
| Russian Federation | 094 | 475 | A |
| Russian Federation | 095 | 331 | В |
| Russian Federation | 095 | 614 | A |
| Russian Federation | 095 | 722 | A |
| Russian Federation | 095 | 478 | В |
| Russian Federation | 096 | 739 | В |
| Russian Federation | 096 | 833 | A |
| Russian Federation | 096 | 755 | A |
| Russian Federation | 096 | 271 | В |
| Russian Federation | 097 | 389 | A |
| Russian Federation | 097 | 668 | В |
| Russian Federation | 097 | 525 | A |
| Russian Federation | 097 | 752 | В |
| Russian Federation | 098 | 842 | A |
| Russian Federation | 098 | 284 | В |
| Russian Federation | 098 | 660 | В |
| Russian Federation | 098 | 826 | A |
| Russian Federation | 099 | 352 | A |
| Russian Federation | 099 | 794 | В |
| Russian Federation | 099 | 143 | В |
| Russian Federation | 099 | 532 | A |
| Russian Federation | 100 | 246 | В |
| Russian Federation | 100 | 135 | A |
| Russian Federation | 100 | 589 | В |
| Russian Federation | 100 | 443 | A |
| Russian Federation | 101 | 211 | A |
| Russian Federation | 101 | 322 | В |
| Russian Federation | 101 | 834 | В |
| Russian Federation | 101 | 446 | A |
| Russian Federation | 102 | 805 | A |




| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 102 | 312 | В |
| Russian Federation | 102 | 966 | A |
| Russian Federation | 102 | 604 | В |
| Russian Federation | 103 | 277 | A |
| Russian Federation | 103 | 511 | В |
| Russian Federation | 103 | 176 | A |
| Russian Federation | 103 | 114 | В |
| Russian Federation | 104 | 915 | В |
| Russian Federation | 104 | 423 | A |
| Russian Federation | 104 | 647 | A |
| Russian Federation | 104 | 550 | В |
| Russian Federation | 105 | 753 | В |
| Russian Federation | 105 | 571 | A |
| Russian Federation | 105 | 634 | A |
| Russian Federation | 105 | 914 | В |
| Russian Federation | 106 | 686 | A |
| Russian Federation | 106 | 113 | В |
| Russian Federation | 106 | 369 | A |
| Russian Federation | 106 | 159 | В |
| Russian Federation | 107 | 852 | В |
| Russian Federation | 107 | 684 | A |
| Russian Federation | 107 | 390 | A |
| Russian Federation | 107 | 622 | В |
| Russian Federation | 108 | 674 | В |
| Russian Federation | 108 | 778 | A |
| Russian Federation | 108 | 947 | A |
| Russian Federation | 108 | 969 | В |
| Russian Federation | 109 | 596 | В |
| Russian Federation | 109 | 751 | A |
| Russian Federation | 109 | 438 | A |
| Russian Federation | 109 | 591 | В |
| Russian Federation | 110 | 666 | В |
| Russian Federation | 110 | 541 | A |
| Russian Federation | 110 | 295 | A |
| Russian Federation | 110 | 106 | В |


07.06.2021



| Country | Block number | Randomization code | Therapy |
|--------------------|--------------|--------------------|---------|
| Russian Federation | 111 | 123 | В |
| Russian Federation | 111 | 100 | A |
| Russian Federation | 111 | 139 | A |
| Russian Federation | 111 | 631 | В |
| Russian Federation | 112 | 302 | A |
| Russian Federation | 112 | 206 | В |
| Russian Federation | 112 | 349 | A |
| Russian Federation | 112 | 420 | В |
| Russian Federation | 113 | 359 | В |
| Russian Federation | 113 | 430 | A |
| Russian Federation | 113 | 797 | В |
| Russian Federation | 113 | 780 | A |
| Russian Federation | 114 | 740 | A |
| Russian Federation | 114 | 457 | В |
| Russian Federation | 114 | 860 | A |
| Russian Federation | 114 | 577 | В |
| Russian Federation | 115 | 606 | В |
| Russian Federation | 115 | 122 | A |
| Russian Federation | 115 | 115 549 | |
| Russian Federation | 115 | 288 | В |

**Therapy A** - Investigational product solution for intravenous and intravenous administration and investigational product film-coated tablets;

**Therapy B** - Placebo 1 solution for intravenous and intravenous administration and Placebo 2 film-coated tablets.

# 6. Main and additional trial parameters to be assessed in the course of the trial

The ITT, mITT and PP populations will be used for efficacy analyses, with the PP population planned to be used as the main population.

The following indicator has been chosen as the **primary efficacy criterion**:

The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the end of therapy vs. baseline (in scores).

The following indicators were selected as **secondary** endpoints:

- The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the end of parenteral therapy vs. baseline (in scores).
- Proportion of disabled patients (mRS score 3 or more) at the end of therapy vs. baseline;
- Proportion of disabled patients (mRS score 3 or more) at the end of parenteral therapy vs. baseline;

07.06.2021



- The magnitude of change in the patient's NIHSS (National Institutes of Health Stroke Scale) score at the end of therapy vs. baseline (in scores).
- The magnitude of change in the patient's NIHSS (National Institutes of Health Stroke Scale) score at the end of parenteral therapy vs. baseline (in scores).
- The magnitude of change in the patient's MoCA cognitive status score at the end of therapy vs. baseline (in scores).
- The magnitude of change in the patient's MoCA cognitive status score at the end of parenteral therapy vs. baseline (in scores).
- The magnitude of change in the patient's Rivermead Mobility Index score at the end of therapy vs. baseline (in scores).
- The magnitude of change in the results of the patient's state assessment by the Rivermead mobility index at the end of the parenteral course of therapy vs. baseline (in scores).
- The magnitude of change in the patient's HADS score at the end of therapy vs. baseline (in scores).
- The magnitude of change in the patient's HADS score at the end of parenteral therapy vs. baseline (in scores).

## The criteria for assessing pharmacodynamic effects are listed below:

- The magnitude of change in the results of assessment of LPO activity (malonic dialdehyde) and AOS indicators (superoxide dismutase, Se-dependent glutathione peroxidase) at the end of therapy vs. baseline;
- The magnitude of change in the results of assessment of LPO activity (malonic dialdehyde) and AOS indicators (superoxide dismutase, Se-dependent glutathione peroxidase) at the end of the parenteral course of therapy vs. baseline;
- The magnitude of change in the results of evaluation of laboratory parameters reflecting ED (Willebrandt factor, endothelin 1, homocysteine) and antihypoxant effect (hypoxia-inducible factor HIF-Iα, lactate, neuron-specific enolase) at the end of therapy vs. baseline;
- The magnitude of change in the results of evaluation of laboratory parameters reflecting ED (Willebrandt factor, endothelin 1, homocysteine) and antihypoxant effect (hypoxia-inducible factor HIF- $1\alpha$ , lactate, neuron-specific enolase) at the end of the parenteral course of therapy vs. baseline.

**Safety and tolerability** will be assessed throughout the trial (from first use of the investigational product/placebo) using the following data:

- 1. AE/SAE reports data,
- 2. Physical examination data, vital signs (BP, HR, respiratory rate, body temperature),
- 3. Indicators of laboratory analyses and instrumental methods of examination.

A conclusion on the safety of the investigational product will be made after statistical evaluation of all AEs, including serious SAEs with at least a possible association with the use of the investigational product.

#### 7. Statistical hypothesis

The trial plans to test the hypothesis of "superiority" of therapy with the investigational product vs. placebo therapy. The following indicator was chosen as the primary efficacy criterion: "The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the



end of therapy (Day 71) vs. baseline (in scores)"

In the case of a superiority trial, the null hypothesis (H0) and the alternative hypothesis (H1) are formulated as follows:

$$H_0$$
:  $\varepsilon = \mu_T - \mu_p \le \delta$ ,  $H_1$ :  $\varepsilon > \delta$ ,  $\delta > 0$ , where

- $\epsilon$  true difference between the value of the primary efficacy index  $(\mu_{\tau})$  in the group of patients taking the investigational product (T) and the value of the primary efficacy index  $(\mu_p)$  in the group of patients taking placebo,
- $\delta$  the boundary of "superiority" of therapy with the investigational product compared to place bo therapy by the primary efficacy indicator.

To prove superiority of therapy with an investigational product compared with placebo therapy, the lower bound of the 95% one-sided confidence interval (CI) for the difference in values of the primary efficacy criterion ( $\mu_{\tau}$  -  $\mu_{p}$ ) must be greater than  $\delta$ , where  $\delta > 0$ , i.e. CI must fall within the interval ( $\delta$ , + $\infty$ ).

#### 8. Estimation of the required sample size

The sample size calculation was based on the results of the Phase III clinical trial of Mexidol® [Multicentre randomized double-blind placebo-controlled parallel-group clinical trial of the safety and efficacy of MEXIDOL® (solution for intravenous and intravenous administration / coated tablets) in long-term sequential therapy in patients with hemispheric ischaemic stroke in the acute and early recovery periods - (EPICA)] dated 30.09.2016.

To calculate the sample size, data from the EPICA clinical trial were used for the ITT population (patients who received the investigational product or placebo at least once), as this population allows us to draw conclusions about the efficacy of the investigational therapy on the population closest to the patient population in real clinical practice.

According to the results of the EPICA clinical trial, the mean value of the change in the mRS score at the end of the course of therapy relative to the baseline level in the group of therapy with the investigational product was (mean (SD)) 278 (0.755) scores, in the placebo group - 1.986 (0.847) scores 2.278 (0.755) scores, in the group of placebo therapy - 1.986 (0.847) scores, the difference (Mexidol® - placebo) is 0.292 scores, 95% confidence interval for the difference (Mexidol® - placebo) is (0.027, 0.556). The "superiority" boundary ( $\delta$ ) was chosen as the lower boundary of the confidence interval constructed for the difference (Mexidol® - placebo). Thus,  $\delta$  = 0.027 scores.

To test the hypothesis of "superiority" of therapy with the investigational product compared with placebo therapy at a significance level of  $\alpha=0.05$  (5%) to ensure power1- $\beta=0.8$  (80%) , the sample size was calculated for the primary efficacy criterion given the parallel design, a 1:1 randomization scheme (i.e., k=1 - the ratio of sample sizes of the groups nT/ ppl.i.e. k=1 - the ratio of sample sizes in the groups  $n_{T}/n_{p}$ ), the expected difference in efficacy between the compared drugs  $\epsilon=0.292$  and with a mixed standard deviation (SD) of the in-group efficacy  $\sigma=0.802$  scores.

The formula [Chow Sh.-Ch., Shao J., Wang H., 2008] was used in the calculation:

$$n_{T}=n_{R}=\frac{(1+1/k) x (z_{a}+z_{\beta}) x \sigma^{2}}{(\varepsilon-\delta)^{2}}$$



where  $z_{\alpha}$  and  $z_{\beta}$  - quantiles of the normal distribution N (0,1) (mean: 0, standard deviation: 1).

The minimum number of patients completing the trial according to the protocol must be at least N=2x 114=228 patients (114 patients per group).

Given the possible attrition of patients in the trial, it is planned to **randomize 304 patients**, of whom at least 228 should complete the trial according to the Protocol.

The trial plans to conduct an interim analysis of the data, based on which a decision will be made whether to end the trial (if the trial objective is met) or to enroll the additional number of patients needed to confirm the efficacy of the drug, followed by pooling of all data for the final analysis.

# 9. Statistical evaluation of efficacy parameters and pharmacodynamic effects

Statistical processing of the data (case report forms of all sites) at the end of the trial will be carried out by staff not involved in the management of the patients participating in the trial, in order to create conditions for independent evaluation of the results obtained. The data will be processed in an electronic database using statistical programmes with the necessary functions (TIBCO® Statistica<sup>TM</sup> v.13 or higher and R v.3.6.2 or higher or other specialised software that determines the appropriate quality of the results obtained).

Descriptive statistics are provided for demographics, baseline values of indices, and values of efficacy and safety indicators at trial visits for the drugs being compared.

Interval (quantitative) data will be described using: arithmetic mean, standard deviation, median, lower (25%) and upper (75%) quartiles, minimum, maximum and coefficient of variation. Categorical (qualitative) data will be described using frequencies, percentages and/or fractions.

The results of quantitative variables evaluation whose distribution follows the law of normal distribution will be presented as  $M\pm SD$ , where M - mean and SD - standard deviation. The results of quantitative variables evaluation whose distribution does not follow the law of normal distribution will be presented as Me [ $Q_1$ ;  $Q_3$ ], where Me - median and  $Q_1$  and  $Q_3$  - lower and upper quartiles.

The Shapiro-Wilk criterion will be applied to select parametric or non-parametric methods of analysis. When testing statistical hypotheses, parametric criteria will be used for indicators that have a normal distribution, and non-parametric criteria will be used for indicators with distribution other than normal. Demographic characteristics and descriptive statistics for baseline indicator values will be presented for the population of all randomized patients.

The primary efficacy variable will be analysed in the PP population (main), and in the ITT and mITT populations (additional). Confirmation of superiority of therapy with Mexidol® solution for intravenous and intramuscular injection, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia) over placebo therapy will be based on the magnitude of change in the patient's mRS (Modified Rankin Scale) scores at the end of the therapy (Day 71) vs. baseline (in scores).

Secondary efficacy and safety endpoints and their changes will be presented using descriptive statistics by visit and therapy group. On trial visits, qualitative (dichotomous) measures will be compared between groups on the basis of Pearson's  $\chi 2$  testor, if the frequency



of a feature in at least one subgroup is 5 or less, Fisher's exact test (or Fisher-Freeman-Galton test for tables of arbitrary dimensionality). Differences with p values of <0.05 will be considered statistically significant.

To compare quantitative data distributed according to the normal distribution law, it is planned to use standard parametric criteria: Student's t-test for dependent/independent samples, analysis of variance (ANOVA) for repeated measures.

It is planned to use standard nonparametric criteria to compare quantitative data distributed according to a law other than normal: Mann-Whitney U-test, Wilcoxon T-test, Friedman's test.

Benjamini-Yekutili correction will be used for multiple statistical hypothesis testing.

A one-sided test will be applied to analyse the primary endpoint and two-sided statistical tests will be applied to analyse all secondary endpoints.

Scatter plots (boxplots) will be presented for all quantitative measures of efficacy and safety. Data whose distribution differs from normal at least at one visit in one of the groups will be presented as median and interquartile range; data whose distribution is normal at all visits will be presented as mean  $\pm$  standard deviation.

Pharmacodynamic effects will be analysed in a subpopulation of patients participating in the evaluation of the pharmacodynamic effects of the investigational therapy.

The resulting data will be analysed using the methods outlined for the application of the efficacy data assessment.

The p-level values < 0.05 will be considered statistically significant.

The trial did not include interim statistical analyses.

The application of methods of statistical analysis of the obtained data will be determined by their nature, type and features of their distribution. The feasibility of using a number of statistical methods will be assessed after the completion of the data set, due to the unknown nature of their distribution, sample homogeneity, etc. During the course of the analysis, it is possible to expand the list of methods used if it is necessary for qualitative data processing.

All data obtained from the trial are subject to analysis. The final analysis of efficacy parameters will be performed after the clinical part of the trial is completed and the electronic database is finalised. If errors are identified in the electronic database prior to finalisation that cannot be resolved after the completion of patient participation in the trial, the statistical analysis of the data will include an analysis of the sensitivity of the resulting parameters to the presence of questionable data.

# 10. Safety analysis

Safety indicators as well as their changes will be presented using descriptive statistics by visit and therapy group. On trial visits, qualitative (dichotomous) measures will be compared between groups on the basis of Pearson's  $\chi^2$  testor, if the frequency of a feature in at least one subgroup is 5 or less, Fisher's exact test (or Fisher-Freeman-Galton test for tables of arbitrary dimensionality).

The dynamics of quantitative safety indicators relative to baseline values will be evaluated and compared with each other using ANOVA analysis of variance with repeated measures. This method allows to simultaneously check the presence of statistically significant dynamics (at least one mean value in one time point differs from the rest), as well as to compare the dynamics and ranges of values of the indicator when receiving the compared preparations. In case of inappropriate use of parametric methods, similar analysis of changes in the distributions of



indicators during therapy will be carried out using non-parametric analogues - Friedman test and Wilcoxon sign rank test, and intergroup comparisons of changes - using the Wilcoxon-Mann-Whitney test.

The number and proportion of patients with reported adverse events after the first dose of the investigational product will be tabulated by therapeutic group. Descriptive statistics for adverse events will also be tabulated, taking into account severity, action taken and outcome.

The safety analyses will descriptively present the values of laboratory parameters as well as their changes from baseline values. In addition, clinically significant and nonsignificant deviations of laboratory values by visit will be tabulated by therapeutic group.

Safety assessment will be carried out based on the analysis of the frequency of occurrence of all adverse events, dynamics of laboratory and instrumental parameters.

AEs are recorded after the first use of the drug until the patient completes the trial and are tracked throughout the trial until they are resolved/stabilised.

Frequency tables with data on discontinuation of therapy or changes in therapy parameters due to AEs will be presented.

Pre- and post-trial data will be compared to assess safety parameters.

All data will be analyzed on the safety population. Regardless of the reason for trial termination, data from all included patients will be included in the safety analyses of the trial therapy.

Adverse event (AE) is any adverse change in the health status of a patient or subject of a clinical trial to whom a medicinal (investigational) product has been administered, regardless of the causal relationship with its use.

**Serious adverse event (SAE)** - any adverse medical event that, regardless of the dose of the medicinal product, has resulted in death, is life threatening, requires hospitalization or its prolongation, has resulted in permanent or significant disability or impairment, is a congenital anomaly or birth defect or other medically significant event.

**Adverse reaction (AR)** - unintentional adverse body reaction associated with the use of a medicinal product/investigational product, suggesting at least a possible relationship with the use of a suspected medicinal product/investigational product.

**Unexpected adverse reaction (UAE)** - an adverse reaction, the nature, severity or outcome of which does not correspond to the information in the current instructions for medical use of the medicinal product or in the investigator's leaflet for an unregistered medicinal product.

**Serious unexpected adverse reaction (SUAR)** - an unexpected adverse reaction that is characterized by features of a SAE.

The parameters of the AE/SAE will be estimated as follows:

#### **Severity of AEs:**

The investigator assesses the severity of an adverse event according to the Common Terminology Criteria for Adverse Events (CTCAE) current version at the time of the trial. If an adverse event cannot be classified according to the CTCAE criteria, the Investigator will select the closest description of the severity of the adverse event from those given in the classification based on personal clinical experience:

- 1. Mild no symptoms or mild symptoms, only clinical or diagnostic follow-up is required; no intervention is indicated;
- 2. Moderate only minimal, localised or non-invasive interventions are indicated; limitation of activities of daily living;


07.06.2021



- 3. Severe severe or clinically significant but not immediately life-threatening; hospitalisation or prolongation of hospitalisation is indicated; loss of ability to work; limitation of self-care in activities of daily living;
- 4. Life-threatening / Disability life-threatening consequences, urgent intervention required;
  - 5. Fatal death associated with an undesirable event.

#### Determination of the relationship of AE to the investigational product:

The investigator should assess the association of the adverse event with the investigational product:

- No clearly and unequivocally related to extraneous causes only, and does not meet the criteria for an unclassifiable, conditional, doubtful, possible, probable or certain relationship.
  - Yes there is a reliable temporal relationship with the use of the medicinal product.

#### Criteria:

- may have been caused by a clinical condition or external factors or other prescribed treatments;
- clear temporal relationship between discontinuation of the investigational product or dose reduction and improvement;
  - resumes upon rechallenge;
  - is consistent with the known nature of the response to the investigational product.

The degree of certainty of causality with the investigational product will be assessed using the WHO scale, taking into account the trial design (multiple administration):

**Definite.** Clinical manifestations of AEs, abnormalities of laboratory parameters occur during the period of drug administration, cannot be explained by the presence of existing diseases and the influence of other factors.

**Probable.** Clinical manifestations of AEs, abnormalities of laboratory parameters are related in time to the use of the drug, unlikely to be related to concomitant diseases or other factors.

**Possible.** Clinical manifestations of AEs, changes in laboratory parameters are related in time to the drug intake, but they can be explained by the presence of concomitant diseases or taking other drugs and the influence of chemical compounds.

**Doubtful.** Clinical manifestations of AEs, changes in laboratory parameters occur in the absence of a clear temporal relationship with the use of the drug; there are other factors (drugs, diseases, chemicals) that may be the cause of their occurrence.

*Conditional.* Clinical manifestations of an AE, abnormalities of laboratory parameters attributed to an AE are difficult to assess. Additional data is needed for evaluation, or the data is currently being analysed.

*Unclassifiable.* Reports of suspected AE cannot be evaluated because there is insufficient information or it is contradictory.

**Foreseeability:** assessed only for AEs considered to be an adverse reaction. An unexpected adverse reaction is an adverse reaction, the nature, severity or outcome of which does not correspond to the information in the current instructions for medical use of the medicinal product or in the investigator's leaflet for an unregistered medicinal product.



The outcome of an AE is assessed as follows:

- Transition to SAE AE resulted in a condition that meets the criteria of seriousness (resulted in death, was life-threatening, required hospitalization of the patient or its prolongation, resulted in permanent or pronounced disability or incapacity, congenital anomalies or malformations, required medical intervention to prevent the development of these conditions. In case of any unexpected suspected transmission of an infectious agent through a medicinal product has occurred);
  - Stabilization of the condition (unchanged condition) the AE has not resolved;
- Recovery with consequences resolution of an AE has occurred, but the patient still has some residual effects;
- Recovery / cessation of an AE without consequences AE has completely resolved with no observable residual effects;
  - Improvement of the condition is a reduction in the severity of an AE;
- Unknown the outcome of an AE is unknown because the patient did not show up for the follow-up examination and attempts to obtain follow-up information were unsuccessful (lost for follow-up).

Clinical laboratory assessments will be presented with descriptive statistics by trial visit indicating changes from baseline. Laboratory abnormalities outside of normal values will be noted. Lists and summary descriptions of clinically significant haematological laboratory abnormalities will be presented. The feasibility of using a number of statistical methods will be assessed after data collection has been completed, as the nature of the data distribution, sample homogeneity, etc. is not known in advance. During the course of the analysis, the list of methods to be used may be modified and supplemented if necessary for the qualitative processing of the data. All deviations from the statistical plan of the survey as well as their causes will be detailed in the statistical report.

Based on the results of the trial, after the final statistical analysis, a conclusion will be made about the efficacy and safety of different dosages in sequential therapy with Mexidol® solution for intravenous and intramuscular administration, 50 mg/ml (RPC PHARMASOFT LLC, Russia) and Mexidol® FORTE 250 film-coated tablets, 250 mg (RPC PHARMASOFT LLC, Russia), vs. placebo. Table templates are provided in the annexes to this statistical plan.

## 11. Patient populations to be analysed

The following population groups will be used for the analyses:

- The ITT (Intent-to-treat) population will include all randomized patients regardless of investigational drug/placebo administration.
- The mITT (modified Intent-to-treat) population will include patients who have completed the full course of therapy, regardless of the presence of Protocol violations/deviations.
- The PP (Per protocol) population will include patients who completed the trial in accordance with the Protocol.
- Subpopulation of patients involved in the evaluation of the pharmacodynamic effects of the investigational therapy: this population will include PP patients with relevant blood test results

The primary population for the evaluation of efficacy criteria, proof of the hypothesis of *Version 1.0 of 12.11.2021* 



superiority of the investigational product therapy over placebo based on the primary efficacy criterion score, will be the PP population. Additionally, efficacy criteria will be analysed in the ITT and mITT populations. Safety parameters will be analysed in the ITT population.

At the stage of statistical data processing, additional analyses of the efficacy and/or safety of investigational product/placebo in subpopulations of patients of different age groups can be performed.

The final report will include data on all patients included in the trial, including those who dropped out at any time without explanation. No missing data will be supplemented.

# 12. Interim analysis

The trial plans to conduct an interim analysis of the data, based on which a decision will be made whether to end the trial (if the trial objective is met) or to enroll the additional number of patients needed to confirm the efficacy of the drug, followed by pooling of all data for the final analysis. The choice of this approach is due to the change in the design of the planned clinical trial, duration of use and dosages of the investigational product compared to the previously conducted clinical trial (EPICA).

In the first phase, an interim analysis of the primary endpoint data will be performed on all randomized patients (304 patients) at the end of the trial:

• If the required power  $\geq$  80% is achieved, a 95% one-sided confidence interval for the difference in values of the primary efficacy criterion ( $\mu_{\tau}$  -  $\mu_{p}$ ) will be used to prove the hypothesis of 'superiority'; the results obtained will be analysed and used to write the final clinical trial report.

If the calculated power is less than 80 per cent, the sample size will be recalculated based on the data obtained after the first stage to achieve a trial power of 80 per cent, using a correction for genus I error  $\alpha$  ( $\alpha$  = 0.0294). A protocol amendment will then be submitted to the Ministry of Health and, once approval is granted, the necessary additional number of patients will be enrolled, followed by pooling of all data for final analysis and writing of the final clinical trial report. A 97.06% one-sided confidence interval for the difference in values of the primary efficacy criterion ( $\mu_{\tau}$  -  $\mu_{p}$ ) constructed from pooled patient data, i.e. obtained from the first and second stage results, using  $\alpha$  = 0.0294, will be used to prove the hypothesis of 'superiority'. The final clinical trial report will be written using data from all patients.

# 13. Table templates

Table 2. Results of assessment of normality of distribution of indicators (template)

| | | Investigational Products | | | | | |
|---|---|---|---|---|---|---|---|
| Indicators Stag | | Mexidol® | | | Placebo | | |
| | | W | P | Distribution | W | P | Distribution |
| Anthropometric parameters | | | | | | | |
| Age | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Height | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Body weight | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |



| BMI V | Stage Visit 0 Visit 0 | W | Mexid<br>P | Distribution normal/other | W | Place<br>P | bo<br>Distribution |
|---|---|---|---|---|---|---|---|
| mRS | | | | | W | P | Distribution |
| mRS | | Eí | | normal/other | | | ~ 10011000001 |
| mRS | | Eí | | | | | normal/other |
| | Visit 0 | Ei | | than normal | | | than normal |
| | Visit 0 | | Efficacy indicators | | | | |
| mRS V | | | | normal/other<br>than normal | | | normal/other<br>than normal |
| mRS I \ | | | | normal/other | | | normal/other |
| l lines | Visit 2 | | | than normal | | | than normal |
| mRS V | Visit 4 | | | normal/other | | | normal/other |
| inics | V 131t ¬ | | | than normal | | | than normal |
| NIHSS V | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| NIHSS V | Visit 2 | | | than normal | | | than normal |
| MILIOO | 71 | | | normal/other | | | normal/other |
| NIHSS | Visit 4 | | | than normal | | | than normal |
| MoCA V | Visit 1 | | | normal/other | | | normal/other |
| | , 1510 1 | | | than normal | | | than normal |
| MoCA V | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| MoCA V | Visit 4 | | | than normal | | | than normal |
| Rivermead V | Visit 1 | | | normal/other | | | normal/other |
| Riverineau | v isit i | | | than normal | | | than normal |
| Rivermead \ | Visit 2 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| Rivermead V | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| HADG A | 7 | | | normal/other | | | normal/other |
| HADS V | Visit 1 | | | than normal | | | than normal |
| HADS V | Visit 2 | | | normal/other | | | normal/other |
| TH IDS | V 151t 2 | | | than normal | | | than normal |
| HADS V | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | Tı | ndicators o | f nharms | acodynamic effect | te | | than normal |
| | | Idicators o | i pharina | normal/other | 1.5 | | normal/other |
| Malonic dialdehyde \ \ | Visit 1 | | | than normal | | | than normal |
| Malonic dialdehyde \ | Visit 2 | | | normal/other | | | normal/other |
| iviaionic dialdenyde | v isit Z | | | than normal | | | than normal |
| Malonic dialdehyde \ | Visit 4 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| Superoxide dismutase \ \ | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Superoxide dismutase \ | Visit 2 | | | normal/other | | | normal/other |



| | | Investigational Products | | | | | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | Mexidol® Pla | | Place | cebo | | |
| | | W | P | Distribution | W | P | Distribution |
| | | | | than normal | | | than normal |
| Superoxide dismutase | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Se-dependent glutathione peroxidase | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Se-dependent glutathione peroxidase | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Se-dependent glutathione peroxidase | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Willebrandt factor | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Willebrandt factor | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Willebrandt factor | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Endothelin 1 | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Endothelin 1 | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Endothelin 1 | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Homocysteine | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Homocysteine | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Homocysteine | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Hypoxia-inducible<br>factor HIF-1α | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Hypoxia-inducible<br>factor HIF-1α | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Hypoxia-inducible<br>factor HIF-Iα | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lactate | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lactate | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lactate | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Neuron-specific enolase | Visit 1 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Neuron-specific enolase | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |


| | | Investigational Products | | | | | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | | Mexid | ol® | | Place | bo |
| | | W | P | Distribution | W | P | Distribution |
| Neuron-specific enolase | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | <u> </u> | Cor | nplete bl | ood count | | | |
| Red blood cells | Visit 0 | | - | normal/other<br>than normal | | | normal/other<br>than normal |
| Red blood cells | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Red blood cells | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haemoglobin | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haemoglobin | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haemoglobin | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haematocrit | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haematocrit | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Haematocrit | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| White blood cells | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| White blood cells | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| White blood cells | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Platelets | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Eosinophils (abs.) | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Eosinophils (abs.) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |



| | | | | Investigation | al Product | S | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | | Mexic | <u> </u> | | Place | bo |
| | | W | P | Distribution | W | P | Distribution |
| Eosinophils (abs.) | Visit 4 | | | normal/other | | | normal/other |
| Losmophiis (aos.) | V 1511 7 | | | than normal | | | than normal |
| Eosinophils (relative) | Visit 0 | | | normal/other | | | normal/other |
| F ( ) | | | | than normal | | | than normal |
| Eosinophils (relative) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| Eosinophils (relative) | Visit 4 | | | than normal | | | than normal |
| | | | | normal/other | | | normal/other |
| Basophils (abs.) | Visit 0 | | | than normal | | | than normal |
| D 1 11 . ( . 1 ) | Minist O | | | normal/other | | | normal/other |
| Basophils (abs.) | Visit 2 | | | than normal | | | than normal |
| Basophils (abs.) | Visit 4 | | | normal/other | | | normal/other |
| Basopinis (aos.) | V 151t ¬ | | | than normal | | | than normal |
| Basophils (relative) | Visit 0 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| Basophils (relative) | Visit 2 | | | normal/other<br>than normal | | | normal/other |
| | | | | normal/other | | | than normal normal/other |
| Basophils (relative) | Visit 4 | | | than normal | | | than normal |
| Bacillary neutrophils | | | | normal/other | | | normal/other |
| (abs.) | Visit 0 | | | than normal | | | than normal |
| Bacillary neutrophils | Minist O | | | normal/other | | | normal/other |
| (abs.) | Visit 2 | | | than normal | | | than normal |
| Bacillary neutrophils | Visit 4 | | | normal/other | | | normal/other |
| (abs.) | V 131t ¬ | | | than normal | | | than normal |
| Bacillary neutrophils | Visit 0 | | | normal/other | | | normal/other |
| (relative) | | | | than normal | | | than normal |
| Bacillary neutrophils (relative) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Bacillary neutrophils | | | | normal/other | | | normal/other |
| (relative) | Visit 4 | | | than normal | | | than normal |
| Segmented neutrophils | | | | normal/other | | | normal/other |
| (abs.) | Visit 0 | | | than normal | | | than normal |
| Segmented neutrophils | V 0 | | | normal/other | | | normal/other |
| (abs.) | Visit 2 | | | than normal | | | than normal |
| Segmented neutrophils | Visit 4 | | | normal/other | | | normal/other |
| (abs.) | v 1511 7 | | | than normal | | | than normal |
| Segmented neutrophils | Visit 0 | | | normal/other | | | normal/other |
| (relative) | | | | than normal | | | than normal |
| Segmented neutrophils | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| (relative) | | | | - | | | |
| Segmented neutrophils (relative) | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| (ICIALIVE) | | | 1 | mun normal | | | man normal |




| | | | | Investigation | nal Product | S | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | | Mexid | ol® | | Place | ebo |
| | | W | P | Distribution | W | P | Distribution |
| Lymphocytes (abs.) | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lymphocytes (abs.) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lymphocytes (abs.) | Visit 4 | | | normal/other<br>than normal | | | normal/other than normal |
| Lymphocytes (relative) | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lymphocytes (relative) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Lymphocytes (relative) | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (abs.) | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (abs.) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (abs.) | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (relative) | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (relative) | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Monocytes (relative) | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| ESR | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| ESR | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| ESR | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | Bioch | nemical b | lood counts | | | |
| Urea | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Urea | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Urea | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Creatinine | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Creatinine | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Creatinine | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |



| | | Investigational Products | | | | | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | | Mexic | lol® | | Place | ebo |
| | | W | P | Distribution | W | P | Distribution |
| Glucose | Visit 0 | | | normal/other | | | normal/other |
| Glucose | V ISIT O | | | than normal | | | than normal |
| Glucose | Visit 2 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| Glucose | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| AST | Visit 0 | | | than normal | | | than normal |
| ACT | Winit 2 | | | normal/other | | | normal/other |
| AST | Visit 2 | | | than normal | | | than normal |
| AST | Visit 4 | | | normal/other | | | normal/other |
| 7101 | V 1510 1 | | | than normal | | | than normal |
| ALT | Visit 0 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| ALT | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| ALT | Visit 4 | | | than normal | | | than normal |
| Total protoin | Visit 0 | | | normal/other | | | normal/other |
| Total protein | VISILU | | | than normal | | | than normal |
| Total protein | Visit 2 | | | normal/other | | | normal/other |
| Total protein | V 1510 2 | | | than normal | | | than normal |
| Total protein | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| Total cholesterol | Visit 0 | | | than normal | | | than normal |
| | | | | normal/other | | | normal/other |
| Total cholesterol | Visit 2 | | | than normal | | | than normal |
| Total cholesterol | Visit 4 | | | normal/other | | | normal/other |
| Total choicsteror | V 1511 4 | | | than normal | | | than normal |
| Triglycerides | Visit 0 | | | normal/other | | | normal/other |
| | | | | than normal | | | than normal |
| Triglycerides | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| | | | | normal/other | | | normal/other |
| Triglycerides | Visit 4 | | | than normal | | | than normal |
| | | l | Vital s | ll | <u> </u> | | |
| ann | <b>37'</b> '. 0 | | 1 | normal/other | | | normal/other |
| SBP | Visit 0 | | | than normal | | | than normal |
| SBP | Visit 2 | | | normal/other | | | normal/other |
| 501 | v 1511 Z | | | than normal | | | than normal |
| SBP | Visit 3 | | | normal/other | | | normal/other |
| | | | 1 | than normal | | | than normal |



| | | | | Investigation | al Product | ts | |
|---|---|---|---|---|---|---|---|
| Indicators | Stage | | Mexid | ol® | | Place | ebo |
| | | W | P | Distribution | W | P | Distribution |
| SBP | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| DBD | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| DBD | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| DBD | Visit 3 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| DBD | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| HR | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| HR | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| HR | Visit 3 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| HR | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| RR | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| RR | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| RR | Visit 3 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| RR | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Body temperature | Visit 0 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Body temperature | Visit 2 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Body temperature | Visit 3 | | | normal/other<br>than normal | | | normal/other<br>than normal |
| Body temperature | Visit 4 | | | normal/other<br>than normal | | | normal/other<br>than normal |



#### Plan for statistical analysis of efficacy and safety parameters

*Table 3. Statistical analysis of the primary endpoint (template)* 

| | | | Mex | kidol® | ı | | | | | Pla | cebo | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MRS scale scores | Visit 0 | Visit 2 | Dynami<br>Visit | | Visit 4 | Dynami<br>Visit | | Visit 0 | Visit 2 | Dynamics to Visit 0 | | Visit 4 | Dynami<br>Visit | |
| | | | Abs. | % | | Abs. | % | | | Abs. | % | | Abs. | % |
| N | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | |
| Qi | | | | | | | | | | | | | | |
| Q3 | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | |
| CV | | | | | | | | | | | | | | |
| | • | | Comp | arison | of drugs (s | statistical te | est <sup>1</sup> ) (p | -value) | • | | | | | - |
| | | Indicator | span diagr | am/ in | dicator sca | tter diagran | n or in | dicator tren | d diagram | | | | | |

Table 4. Outcome of primary endpoint analysis (template)

| Primary endpoint Mexidol® vs. Placebo |
|---------------------------------------|
|---------------------------------------|

<sup>&</sup>lt;sup>1</sup> T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator *Version 1.0 of 12.11.2021* 



#### Plan for statistical analysis of efficacy and safety parameters

| | Difference in means | 95% CI <sup>2</sup> lower limit | 95% CI,<br>upper limit | Power, % <sup>3</sup> | Superiority is confirmed <sup>4</sup> |
|---|---|---|---|---|---|
| The magnitude of change in the patient's mRS (Modified Rankin Scale) score at the end of therapy vs. baseline (in scores). | | | | | |

Table 5. Statistical analysis of the NIHSS scale (template)

| | | | Mex | kidol® | 1 | | | Placebo | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| NIHSS scores | Visit 0 | Visit 2 | Dynami<br>Visit | | Visit 4 | Dynami<br>Visit | | Visit 0 | Visit 2 | Dynami<br>Visit | | Visit 4 | Dynami<br>Visit | |
| | | | Abs. | % | | Abs. | % | | | Abs. | % | | Abs. | <b>%</b> |
| N | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | |
| Qi | | | | | | | | | | | | | | |
| Q3 | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | |
| CV | | | | | | | | | | | | | | |

 $<sup>^2</sup>$  Or "97.06% CI" for Stage 2


Protocol-Specific Version for Protocol #PHS-APIS-004-MEX-SOL-TAV. version 1.3 dated

<sup>&</sup>lt;sup>3</sup> Applicable for Stage 1 only

<sup>&</sup>lt;sup>4</sup> According to the Clinical Trial Protocol, a conclusion of superiority can be made if the upper bound of the two-sided 95% confidence interval for the difference in mean changes in the mean deviation (MD) of Mexidol® compared to placebo is greater than the margin of superiority of investigational product therapy vs. placebo therapy.



| Comparison of drugs (statistical test <sup>5</sup> ) (p-value) |
|---|
| Indicator span diagram/ indicator scatter diagram or indicator trend diagram |

*Table 6. Statistical analysis of secondary endpoints (quantitative data, template)* 

| | | | Mex | idol® | | | | | | Pla | cebo | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Indicator <sup>6</sup> | Visit1 | Visit 2 | Dynamics to<br>Visit 0 | | Visit 4 | _ | Dynamics to Visit 0 | | Visit 2 | Dynamics to Visit 0 | | Visit 4 | Dynamics to<br>Visit 0 |
| | | | Abs. | . % Abs. % | | | Abs. % | % | | Abs. | % | | |
| N | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | |
| Qi | | | | | | | | | | | | | |
| Q3 | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | |
| CV | | | | | | | | | | | | | |
| | Comparison of drugs (statistical test <sup>7</sup> ) (p-value) | | | | | | | | | | | | |
| | Indicator span diagram/ indicator scatter diagram or indicator trend diagram | | | | | | | | | | | | |

<sup>&</sup>lt;sup>5</sup> T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator

<sup>&</sup>lt;sup>6</sup> MoCA and HADS scales, Rivermead index scores

<sup>&</sup>lt;sup>7</sup> T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator *Version 1.0 of 12.11.2021* 



Table 7. Statistical analysis of pharmacodynamic effect indicators (template)

| | | | Mex | idol® | | | | | | Pla | cebo | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Indicator <sup>8</sup> | Visit 1 | Visit 1 Visit 2 | Visit 2 Dynamics Visit 0 | | Visit 4 | Dynamics to<br>Visit 0 | | Visit 1 | Visit 2 | Dynamics to Visit 0 | | Visit 4 | Dynamics to<br>Visit 0 | |
| | | | Abs. | % | | Abs. | % | | | Abs. | % | | Abs. | % |
| N | | | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | | | |
| Median | | | | | | | | | | | | | | |
| Min | | | | | | | | | | | | | | |
| Max | | | | | | | | | | | | | | |
| Qi | | | | | | | | | | | | | | |
| Q3 | | | | | | | | | | | | | | |
| SD | | | | | | | | | | | | | | |
| CV | | | | | | | | | | | | | | |
| | Comparison of drugs (statistical test <sup>9</sup> ) (p-value) | | | | | | | | | | | | | |
| | Indicator span diagram/ indicator scatter diagram or indicator trend diagram | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>8</sup> Indicators of LPO activity (malonic dialdehyde) and AOS indicators (superoxide dismutase, Se-dependent glutathione peroxidase), as well as indicators reflecting ED (Willebrandt factor, endothelin 1, homocysteine) and antihypoxant action (hypoxia-inducible factor HIF-1α, lactate, neuron-specific enolase).

<sup>&</sup>lt;sup>9</sup> T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator *Version 1.0 of 12.11.2021* 



Table 8. Statistical analysis of the proportion of disabled patients (template)

| | | Vis | it 2 | Visit | 4 |
|---|---|---|---|---|---|
| Percentage of disabled p | oatients | Mexidol® | Placebo | Mexidol® | Placebo |
| Observed | Abs. | | | | |
| Observed | % | | | | |
| | Abs. | | | | |
| Not observed | % | | | | |
| | % | | | | |
| Compariso | Comparison of groups (statistical criterion <sup>10</sup> ) | | | | |

Table 9. Statistical analysis of safety indicators (quantitative data, template)

| | | <b>Mexidol</b> ® | | | | | | Placebo | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Safety<br>indicator <sup>11</sup> | Visit 0 | Visit 2 | Visit | Dynami<br>Visit | | Visit 0 | Visit 2 | Visit 4 | Dynami<br>Visit | |
| | | 2 | 4 | Abs. | % | U | | | Abs. | % |
| N | | | | | | | | | | |
| Mean | | | | | | | | | | |
| Median | | | | | | | | | | |
| Min | | | | | | | | | | |
| Max | | | | | | | | | | |
| Qi | | | | | | | | | | |
| Q3 | | | | | | | | | | |
| SD | | | | | | | | | | |
| CV | | | | | | | | | | |
| | Comparison of drugs (statistical test <sup>12</sup> ) (p-value) | | | | | | | | | |
| Indicator | span dia | agram/ | indicato | or scatter | diagra | m or in | dicator | trend dia | agram | |

Table 10. Statistical analysis of vital signs (quantitative data, template)

| · · |
|-----|
|-----|

<sup>&</sup>lt;sup>10</sup> Pearson 's χ2 criterion or Fisher's exact test

<sup>&</sup>lt;sup>11</sup> Clinical and biochemical blood counts.

 $<sup>^{12}</sup>$  T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator  $Version\ 1.0\ of\ 12.11.2021$ 



| indicator <sup>13</sup> | Visit 0 | Visit 2 | Visit 3 | Visit 4 | Dynan<br>to Vis | | Visit 0 | Visit 2 | Visit 3 | Visit 4 | Dynan<br>to Visi | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | U | 2 | 3 | 4 | Abs. | % | U | 4 | 3 | + | Abs. | % |
| N | | | | | | | | | | | | |
| Mean | | | | | | | | | | | | |
| Median | | | | | | | | | | | | |
| Min | | | | | | | | | | | | |
| Max | | | | | | | | | | | | |
| Qi | | | | | | | | | | | | |
| Q3 | | | | | | | | | | | | |
| SD | | | | | | | | | | | | |
| CV | | | | | | | | | | | | |
| | Comparison of drugs (statistical test <sup>14</sup> ) (p-value) | | | | | | | | | | | |
| Indica | tor spai | n diagr | am/ in | dicato | r scatter | diag | ram or | indica | tor trer | nd diag | ram | |

Table 11. Safety performance assessment results: repeated measures analysis of variance (template)

| Safety<br>Indicator/Investigational<br>Product | SS | DF | MS | F | р |
|------------------------------------------------|----|----|----|---|---|
| Intercept | | | | | |
| Investigational Product | | | | | |
| Error | | | | | |
| Visit | | | | | |
| Visit*Dru | | | | | |
| Error | | | | | |

Table 12.Results of safety indicators assessment: non-parametric repeated measures analysis of variance (Friedman test, template)

| Investigational Product | | | | | |
|-------------------------|--------------|--------------|------|----|---|
| Indicator | | | | | |
| Visit | Average rank | Sum of ranks | Mean | SD | р |
| Visit 1 | | | | | |
| ••• | | | | | |

<sup>&</sup>lt;sup>13</sup> SBP, DBP, HR, RR, body temperature.

<sup>&</sup>lt;sup>14</sup> T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator Version 1.0 of 12.11.2021



Table 13. Frequency analysis of safety performance outcome assessment (template)

| | | | | ) | Placebo | |
|---|---|---|---|---|---|---|
| Investigational Pro | Visit 0 | Visit 2 | Visit 4 | Visit 0 | Visit 2 | Visit 4 |
| | Inc | dicator 1 | _ | • | | |
| Name of | Abs. | | | | | |
| Normal | % | | | | | |
| | Abs. | | | | | |
| Deviation | % | | | | | |
| | % | | | | | |
| Comp | parison of grou | ups (stati | stical cri | terion <sup>15</sup> ) | ) | |
| | p-level | | | | | |
| | Inc | dicator 2 | 2 | | | |
| | | ••• | | | | |

Table 14. Frequency analysis of the safety outcome measure score (clinical significance, template)

| | | M | Mexidol® | | | Placebo |
|---|---|---|---|---|---|---|
| Investigational Produc | Visit 0 | Visit 2 | Visit 4 | Visit 0 | Visit 2 | Visit 4 |
| | Indica | tor 1 | | | | |
| Deviation is clinically significant | Abs. | | | | | |
| | % | | | | | |
| D | Abs. | | | | | |
| Deviation is clinically insignificant | % | | | | | |
| msignificant | % | | | | | |
| Comparison of groups (statistical criterion <sup>16</sup> ) | | | | | | |
| p-le | p-level | | | | | |
| | Indica | tor 2 | | | | |

<sup>&</sup>lt;sup>15</sup> Pearson 's γ2 criterion or Fisher's exact test


<sup>&</sup>lt;sup>16</sup> Pearson 's  $\chi^2$  criterion or Fisher's exact test



Table 15. Statistical analysis of ECG (template)

| | | | | Mexidol® | | | |
|---|---|---|---|---|---|---|---|
| Investigational Proc | luct | Visit 0 | Visit 2 | Visit 4 | Visit 0 | Visit 2 | Visit 4 |
| No | Abs. | | | | | | |
| Normal | % | | | | | | |
| | Abs. | | | | | | |
| Deviation | % | | | | | | |
| | % | | | | | | |
| Comp | arison of gro | ups (stati | stical crit | terion <sup>17</sup> ) | | | |
| | p-level | | | | | | |

Table 16. Statistical analysis of physical examination parameters (outcome measure, template)

| | | | Mexidol® | | | | Plac | ebo | |
|---|---|---|---|---|---|---|---|---|---|
| Investigational Product | | Visit 0 | Visit 2 | Visit 3 | Visit 4 | Visit 0 | Visit 2 | Visit 3 | Visit 4 |
| Indicator 1 | | | | | | | | | |
| Normal | Abs. | | | | | | | | |
| Normai | % | | | | | | | | |
| | Abs. | | | | | | | | |
| Deviation | % | | | | | | | | |
| | % | | | | | | | | |
| C | Comparison of groups (statistical criterion <sup>18</sup> ) | | | | | | | | |
| p-level | | | | | | | | | |
| | Indicator 2 | | | | | | | | |
| | | | ••• | | | | | | |

Table 17. Distribution of patients by ender (template)

| Gender | | <b>Mexidol</b> ® | Placebo |
|--------|------|------------------|---------|
| Female | Abs. | | |
| remale | % | | |
| Male | Abs. | | |

<sup>&</sup>lt;sup>17</sup> Pearson 's γ2 criterion or Fisher's exact test


<sup>&</sup>lt;sup>18</sup> Pearson 's  $\chi^2$  criterion or Fisher's exact test



| % | |
|---------------------|-------------------------|
| Differences between | Pearson 's χ2 criterion |
| groups | |

#### Table 18. Baseline patient characteristics (template)

| Indicator <sup>19</sup> | Mexidol® | Placebo |
|---|---|---|
| N | | |
| Mean | | |
| Median | | |
| Min | | |
| Max | | |
| Qi | | |
| Q3 | | |
| SD | | |
| CV | | |
| Comparison of groups | Statistic | cal criterion <sup>20</sup> , p-value |
| I | Range diagram | Scatter diagram |

#### Table 19. Total number of AEs (template)

| AE | After administration of | |
|---------------------------------------|-------------------------|---------|
| AE | Mexidol® | Placebo |
| Total number of AEs | | |
| Number of noticets with detected A.C. | Abs. | |
| Number of patients with detected AEs | % | |

#### Table 20. Relative risk of AEs (template)

| Presence of adverse events in patients | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Abs. | | | |
| Identified | % | | |
| Not identified | Abs. | | |
| Not identified | % | | |
| Differences between preparations | | Pearson 's χ2 criterion or Fisher's exact test | |
| Relative risk of AEs [95% CI] | | | |

Age, height, body weight or BMI
 T-test for independent samples or Mann-Whitney test depending on the type of distribution of the indicator Version 1.0 of 12.11.2021



Table 21. Analysing the distribution of AEs by severity (template)

| Severity | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Mild | Abs. | | |
| Milia | % | | |
| Moderate | Abs. | | |
| Moderate | % | | |
| Severe | Abs. | | |
| Severe | % | | |
| Life-threatening/ | Abs. | | |
| Disability to work | % | | |
| Fatal | Abs. | | |
| ratai | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or Fisher's exact test | p-value |

Table 22. Relationship of AEs to investigational product (template)

| The association of the adverse event with the investigational drug | | Investigational Product | |
|---|---|---|---|
| | | <b>Mexidol</b> ® | Placebo |
| Vac | Abs. | | |
| Yes | % | | |
| No | Abs. | | |
| No | % | | |
| Differences between preparations | | Pearson 's χ2 criterion or<br>Fisher's exact test | p-value |

Table 23: Analysis of the distribution of AEs by administration of the Investigational Product (template)

| Relationship to Investigational Product administration | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Definite. | Abs. | | |
| Definite. | % | | |
| Probable. | Abs. | | |
| Probable. | % | | |
| Possible. | Abs. | | |
| | % | | |
| Doubtful. | Abs. | | |


 ${\it Protocol-Specific Version for Protocol \#PHS-}$ 



| | % | | |
|---|---|---|---|
| Conditional. | Abs. | | |
| | % | | |
| Unclassifiable. | Abs. | | |
| Officiassifiable. | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or<br>Fisher's exact test | p-value |

Table 24. Analysis of the distribution of AEs by foreseeability (template)

| Expectancy | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Evmontod | Abs. | | |
| Expected | % | | |
| I In average d | Abs. | | |
| Unexpected | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or Fisher's exact test | p-value |

Table 25. Analysis of AR distribution (template)

| AE | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| A D | Abs. | | |
| AR | % | | |
| N. A.D. | Abs. | | |
| Not an AR | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or<br>Fisher's exact test | p-value |

Table 26. Analysis of the distribution of AEs by seriousness (template)

| Seriousness | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Serious | Abs. | | |
| Serious | % | | |
| Nagagiana | Abs. | | |
| Nonserious | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or<br>Fisher's exact test | p-value |

Table 27. Analysing the distribution of AEs by actions taken (template)



| Actions taken | Investigational Product | | |
|---|---|---|---|
| Actions taken | Mexidol® | Placebo | |
| No action was taken | | | |
| Other (specific actions taken will be indicated) | | | |
| Inter-group differences | | Pearson 's χ2 criterion or Fisher's exact test | p-value |

Table 28. Analysis of the distribution of AEs by outcome (template)

| Outcome | | Investigational Product | |
|---|---|---|---|
| | | Mexidol® | Placebo |
| Transition to SAE | Abs. | | |
| Transition to SAE | % | | |
| Stabilization of the | Abs. | | |
| condition (no change in condition): | % | | |
| Recovery with | Abs. | | |
| consequences | % | | |
| Recovery/termination of | Abs. | | |
| an AE without consequences: | % | | |
| Immerced condition | Abs. | | |
| Improved condition | % | | |
| Unknown: | Abs. | | |
| | % | | |
| Inter-group differences | | Pearson 's χ2 criterion or Fisher's exact test | p-value |



Table 29. Summary table of the incidence of reported AEs in the group taking Mexidol by severity with randomization numbers of patients (N=) (template)

| AE/code, PT according to<br>MedDRA version | Mild | Mild AE Me | | Medium AE Mod | | Moderate AE | | Life-threatening AE | | Fatal AE | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA version | R | UR | R | UR | R | UR | R | UR | R | UR | R | UR | R+UR |

Table 30. Summary table of the incidence of reported AEs in the group taking placebo by severity with randomization numbers of patients (N=) (template)

| Adverse event/code, PT level | | Mild AE Med | | Medium AE Moderate | | ate AE | AE Life-threatening AE | | Fatal AE | | Total | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| according to MedDRA version | R | UR | R | UR | R | UR | R | UR | R | UR | R | UR | R+UR |

Table 31. Summary table of the incidence of AEs after taking each Investigational Product (template)

| A dyrange expent/gode DT level according to ModDDA yengion | Mexido | ol N= | Place | ebo N= | P-value (Statistical |
|---|---|---|---|---|---|
| Adverse event/code, PT level according to MedDRA version | n | % | n | % | criterion) |



### Plan for statistical analysis of efficacy and safety parameters

#### *Table 32. List of all adverse events for each patient (template)*

| Site<br>numbe<br>r | Randomizatio<br>n number, full<br>name | Demographi<br>c data | AE/code,<br>PT<br>accordin<br>g to<br>MedDRA<br>version | AE<br>onse | Severit<br>y | Seriousnes<br>s | Relationshi<br>p | rolatio | in relation to<br>the | t thorany | Date<br>the AE<br>resolve<br>d | l I |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Age, years | | | | | | | | | | |
| | | gender | | | | | | | | | | |
| | | Weight, | | | | | | | | | | |
| | | kg | | | | | | | | | | |
| | | Height, | | | | | | | | | | |
| | | cm | | | | | | | | | | |
| | | race | | | | | | | | | | |

# Table 33. MedDRA version classification of AEs (template)

| Randomization number, initials | AE | MedDRA AE code,<br>SOC level | MedDRA AE term,<br>SOC level | MedDRA AE code, PT<br>level | MedDRA AE term, PT<br>level |
|---|---|---|---|---|---|



#### Plan for statistical analysis of efficacy and safety parameters

Table 34. Summary table of the incidence of reported SAEs in the group taking Mexidol by severity with randomization numbers of patients (N=) (template)

| Adverse event/code, PT level | | Mild AE Medium A | | ım AE | E Moderate AE | | Life-threatening<br>AE | | Fatal AE | | Total | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| according to MedDRA version | R | UR | R | UR | R | UR | R | UR | R | UR | R | UR | R+UR |

Table 35. Summary table of the incidence of reported SAEs in the placebo group by grade with randomization numbers of patients (N=) (template)

| Adverse event/code, PT level | Mild | AE | Medium AE | | Moderate AE | | Life-threatening<br>AE | | Fatal AE | | Total | | Total |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| according to MedDRA version | R | UR | R | UR | R | UR | R | UR | R | UR | R | UR | R+UR |

Table 36. Summary table of the incidence of SAEs after taking each investigational product (template)



### Plan for statistical analysis of efficacy and safety parameters

| | Mexid | ol® | Plac | ebo | D value (Statistical |
|---|---|---|---|---|---|
| Adverse event/code, PT level according to MedDRA version | N= | | N | | P-value (Statistical criterion) |
| | n | % | n | % | Ci itelion) |

Table 37. List of all serious adverse events for each patient (template)

| Site<br>numbe<br>r | Randomizatio<br>n number, full<br>name | Dama awan bi | SAE/code<br>, PT<br>according<br>to<br>MedDRA<br>version | Severit<br>y | Seriousnes<br>s | Relationshi<br>p | Actions taken in relation to the patient | in relation to<br>the | t thorany | Date<br>the AE<br>resolve<br>d |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Age, years | | | | | | | | |
| | | gender | | | | | | | | |
| | | Weight, | | | | | | | | |
| | | kg | | | | | | | | |
| | | Height, | | | | | | | | |
| | | cm | | | | | | | | |
| | | race | | | | | | | | |

Table 38. MedDRA version classification of SAEs (template)





| Randomization number, initials | SAE | SAE MedDRA code,<br>SOC level | SAE MedDRA term,<br>SOC level | SAE MedDRA code,<br>PT level | SAE MedDRA term,<br>PT level |
|---|---|---|---|---|---|